CLINICAL TRIAL: NCT04896983
Title: National Survey of Mental Health in the Second Year After COVID-19 Outbreak: Multilevel Analysis of Individual and Societal Factors
Brief Title: National Survey of Mental Health After COVID-19 Outbreak
Acronym: CoV2SoulRS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Belgrade (Other)
Collaborators: University of Novi Sad (Other)
Responsible Party: Principal Investigator, Nadja P Maric, Principal Research Fellow & Professor, University of Belgrade
Other Study IDs: #7528289; #7528289 COVID-19 CoV2Soul.RS (Other Grant/Funding Number: Science Fund of the Republic of Serbia)
Record Dates: First submitted 2021-05-12; First posted 2021-05-21 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Mental Health Impairment
Keywords: COVID-19; Prevalence; Mental health disorders; Stress; Personality; Multilevel modelling; National survey; Quality of life
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Serbian national survey - acronym CoV2Soul.RS - has been launched to document mental health (MH) status and understand needs of the population in relation to the prolonged global public health crisis.

This cross-sectional study will collect a representative national sample (18-65 years) by multi-stage probabilistic household sampling method. Trained staff will conduct face-to-face diagnostic interviews (M.I.N.I.). Battery of self-report instruments will be used to measure quality of Life (QoL), level of distress, and associated protective and harmful psychological and societal factors. The investigators aim to assess prevalence rates of MH disorders and associated QoL in the nationally representative sample, to explore how MH conditions and QoL vary with respect to socio-demographic variables, personality, health status and traumatic events during pandemics, and to find how these relationships depend on societal factors characterising municipalities in which they live. Moreover, this study will address perception of pandemic consequences and associated distress in relation to personality and different types of possible mediators. The prevalence rates of MH disorders will be calculated as percentages of participants with a positive diagnosis. The hierarchical structure of the data will be analyzed using Multilevel Random Coefficient Modeling,

CoV2Soul.RS will contribute to an international evidence base about prevalence rates of psychiatric conditions during different phases of the pandemic in different regions and will identify protective and harmful psychological and societal factors for MH and QoL.

ELIGIBILITY:
Inclusion criteria:

* Age between 18 and 65 years
* Speaks Serbian fluently
* Able to give informed consent

Exclusion criteria:

* Cognitive impairment leading to a disability to understand questions
* Severe neurological impairment
* People with impaired hearing and deaf persons

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The sample will be collected via multi-stage probabilistic household sampling (face-to-face, computer-assisted, or paper-pencil method). The first stage includes a random sampling of municipalities as clusters, while the second stage includes a random sampling of local communities in each municipality. Municipalities and local communities are sampled from four regions (Capital Belgrade and suburbs, Vojvodina, West, and Southeast Serbia) based on the random selection from the database created by the Serbian Institute of Statistics (database includes information on the name of the settlement, municipality, region, and the number of inhabitants). The third, final stage, deals with the selection of the respondents using a random walk technique.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Prevalence of MH disorders | Up to 24 weeks
  Prevalence of 16 most common mental health disorders assessed by M.I.N.I 7.0.2, Standard Adult version (Sheehan et al, 1998) / Seven categories of MH conditions: (1) Mood disorders (Major depressive episode, Manic episode and Hypomanic episode); (2) Psychotic disorders; (3) Anxiety disorders (panic disorder, agoraphobia, social phobia, and generalized anxiety disorder); (4) Obsessive-compulsive disorder; (5) Trauma-related disorders (Post-traumatic stress disorder); (6) Eating disorders, and (7) Substance-related and addictive disorders.
Severity of depressive symptoms | Up to 24 weeks
  Depressive symptom severity will be measured by Patient Health Questionnaire - PHQ-9 (Kroenke et al., 2001); Score range 0-27 (higher scores inidicate more severe symptoms)
Severity of anxiety symptoms | Up to 24 weeks
  Anxiety symptom severity will be measured by General Anxiety Disorder - GAD-7 (Spitzer et al., 2006). Score range 0-21 (higher scores indicate more severe symptoms)
Intensity of the pandemic-related stress | Up to 24 weeks
  Covid Stress Scale (Taylor et al., 2020) will be used. Score range 0-4. Higher score means worse pandemic-related psychological problems.
Perception of COVID-19 pandemic consequences | Up to 24 weeks
  Perception of the pandemic consequences on various aspects of life will be measured using 6 items, allowing for positive Covid-19 related consequences. Score range 1-5.
  Lower score means more negative perception of the pandemic consequences.
Quality of life in relation to different MH conditions | Up to 24 weeks
  QoL assumes focusing on satisfaction with life as a whole (to be assessed by Manchester Short Assessment of Quality of Life - MANSA (Priebe et al., 1999). Score range: 1-7. Higher score means better QoL.
Quality of life in general | Up to 24 weeks
  Short Form survey scale - SF-12 (Ware et al., 1996) - to measure two specific QoL outcomes: 1) physical health-related quality of life (scores range: 6-20), and b) mental health-related quality of life (scores range: 6-27). Higher score means better QoL.

CONTACTS AND LOCATIONS:
Locations (3):
- Serbia (3):
  - Faculty of Medicine, University of Belgrade, Belgrade
  - Faculty of Philosophy, University of Belgrade, Belgrade
  - Faculty of Philosophy, University of Novi Sad, Novi Sad

IPD SHARING:
Plan to Share IPD: Yes
Collected data will be completely anonymized and used in subsequent analyses at the group level. Anonymized dataset will be uploaded to a repository following all good scientific practices.

REFERENCES:
- [Background] Taylor S, Landry CA, Paluszek MM, Fergus TA, McKay D, Asmundson GJG. Development and initial validation of the COVID Stress Scales. J Anxiety Disord. 2020 May;72:102232. doi: 10.1016/j.janxdis.2020.102232. Epub 2020 May 4. PMID 32408047
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Priebe S, Huxley P, Knight S, Evans S. Application and results of the Manchester Short Assessment of Quality of Life (MANSA). Int J Soc Psychiatry. 1999 Spring;45(1):7-12. doi: 10.1177/002076409904500102. PMID 10443245
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Derived] Maric NP, Lazarevic LB, Mihic L, Pejovic Milovancevic M, Terzic Z, Toskovic O, Todorovic J, Vukovic O, Knezevic G. Mental health in the second year of the COVID-19 pandemic: protocol for a nationally representative multilevel survey in Serbia. BMJ Open. 2021 Sep 21;11(9):e053835. doi: 10.1136/bmjopen-2021-053835. PMID 34548371
- See also: Web-site — http://cov2soul.rs